CLINICAL TRIAL: NCT00641147
Title: Curcumin for Treatment of Intestinal Adenomas in Familial Adenomatous Polyposis (FAP)
Brief Title: Curcumin in Treating Patients With Familial Adenomatous Polyposis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2013-00536; NCI-2013-00536 (Other: NCI); CDR0000592794 (Other: Clinical Trial Reporting Program); NA_00011821 (Other: Johns Hopkins University IRB); 1R01CA134620 (NIH); R01CA134620 (NIH); P30CA006973 (NIH)
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Familial Adenomatous Polyposis
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (curcumin) (Experimental): Patients receive curcumin PO BID for 12 months. Laboratory Biomarker Analysis
  Interventions: Drug: Curcumin; Other: Laboratory Biomarker Analysis
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO BID for 12 months. Laboratory Biomarker Analysis
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo

INTERVENTIONS:
Drug: Curcumin — Given PO
  Other Names: C.I. 75300; C.I. Natural Yellow 3; Diferuloylmethane; Turmeric Yellow
  Arms: Arm I (curcumin)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; sham therapy
  Arms: Arm II (placebo)

SUMMARY:
This randomized phase II trial studies curcumin in treating patients with familial adenomatous polyposis. Curcumin may prevent colorectal cancer in patients with a history of rectal polyps or colorectal neoplasia.

DETAILED DESCRIPTION:
Specific Aims:

I. To determine in a randomized, double-blinded, placebo-controlled study the tolerability and effectiveness of curcumin to regress intestinal adenomas by measuring duodenal and colorectal/ileal polyp number, and polyp size in familial adenomatous polyposis patients with intact colons, ileorectal anastomosis surgery, or ileo-anal pullthrough (reservoir) surgery.

II. To measure markers of cell proliferation including colorectal mucosal levels of ornithine decarboxylase (ODC), polyamines, mucosal deoxyribonucleic acid (DNA) methylation, proliferative index (Ki67 antiproliferative cell nuclear antibody), apoptosis index, vascular density, mucosal prostaglandin, leukotriene levels, and activation of the nuclear factor kappa B (NFKB), and v-akt murine thymoma viral oncogene homolog 1 (Akt) survival pathways.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive curcumin orally (PO) twice daily (BID) for 12 months.

Arm II: Patients receive placebo PO BID for 12 months.

After completion of study treatment, patients are followed up at 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with familial adenomatous polyposis who have undergone subtotal colectomy with ileorectal anastomosis, total colectomy with ileo-anal pull through (reservoir), and patients with intact colons with 5 or more adenomas in the rectum-sigmoid or reservoir
* Patients with familial adenomatous polyposis (FAP) and duodenal adenomatous polyposis without current lower tract adenomatous polyposis i.e. status/post (s/p) ileostomy

Exclusion Criteria:

* Female patients of childbearing age not on effective birth control
* Pregnant women
* White blood cell count (WBC) < 3500/ml
* Platelet count < 100,000/ml
* Blood urea nitrogen (BUN) > 25mg%
* Creatinine > 1.5mg%
* Patients unable to stop non-steroidal anti-inflammatory drugs (NSAIDs), aspirin, curcumin, tumeric, calcium, vitamin D, green tea, or polyphenol E supplements for the duration of the trial
* Malignancy other than nonmelanoma skin cancer
* Active bacterial infection
* Patients with symptoms of active gastroesophageal reflux disease (GERD) (symptomatic despite medication or current erosive esophagitis on endoscopy)
* Patients with a history of peptic ulcer disease
* Patients on warfarin or plavix

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Giardiello, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (2):
- Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland, United States
- University of Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cruz-Correa M, Hylind LM, Marrero JH, Zahurak ML, Murray-Stewart T, Casero RA Jr, Montgomery EA, Iacobuzio-Donahue C, Brosens LA, Offerhaus GJ, Umar A, Rodriguez LM, Giardiello FM. Efficacy and Safety of Curcumin in Treatment of Intestinal Adenomas in Patients With Familial Adenomatous Polyposis. Gastroenterology. 2018 Sep;155(3):668-673. doi: 10.1053/j.gastro.2018.05.031. Epub 2018 May 23. PMID 29802852

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at the Johns Hopkins Hospital and the University of Puerto Rico Hospital.
Groups:
- Arm I (Curcumin): Patients receive curcumin by mouth (PO) twice a day (BID) for 12 months.
  Curcumin: Given PO
- Arm II (Placebo): Patients receive placebo PO BID for 12 months.
  Placebo: Given PO
Period: Completed 4 Months.
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Started | 21 | 23
Completed | 19 | 23
Not Completed | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Completed 8 Months.
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Started | 19 | 23
Completed | 16 | 21
Not Completed | 3 | 2
Not completed — Physician Decision | 2 | 1
Not completed — non compliance | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Completed 12 Months.
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Started | 16 | 21
Completed | 15 | 19
Not Completed | 1 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Completed 16 Months.
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Started | 15 | 19
Completed | 13 | 19
Not Completed | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Curcumin): Patients receive curcumin PO BID for 12 months.
  Curcumin: Given PO
- Total: Total of all reporting groups
Arm/Group | Arm I (Curcumin) | Arm II (Placebo) | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (15.4) | 38.7 (15.0) | 41.5 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 22
  Not Hispanic or Latino | 10 | 12 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 21 | 22 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline number of polyps [Mean (Standard Deviation); unit: polyps] | 23.3 (19.7) | 18.7 (13.1) | 20.9 (16.6)
Baseline size of polyps in mm [Mean (Standard Deviation); unit: polyps] | 3.1 (1.7) | 2.3 (0.6) | 2.6 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Polyp Number
Description: Average number of polyps in the placebo arm at the end of the study is compared to the average in the curcumin arm
Time Frame: Up to 12 months
Measure: Mean (95% Confidence Interval); unit: polyps
Groups:
- Arm I (Curcumin): Patients receive curcumin 3.0 grams PO BID for 12 months.
  Curcumin: Given PO
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 16 | 21
polyps | 22.6 [12.1 to 33.1] | 18.6 [9.3 to 27.8]
Statistical Analysis 1: Comparison: Arm I (Curcumin) vs Arm II (Placebo); Test type: Superiority; p = 0.58, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm I (Curcumin) vs Arm II (Placebo); Test type: Superiority; p = 0.57, ANCOVA

2. Secondary Outcome: Mean Polyp Size in mm
Description: Mean size of the 5 largest polyps
Time Frame: Up to 12 months
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 16 | 21
mm | 2.3 [1.6 to 3.0] | 2.1 [1.5 to 2.7]
Statistical Analysis 1: Comparison: Arm I (Curcumin) vs Arm II (Placebo); Test type: Superiority; p = 0.76, t-test, 2 sided

3. Secondary Outcome: Number of Participants With a Decrease in Polyp Burden at 12 Months
Description: The polyp burden as evaluated by video tape review. Polyp burden at 12 months compared to time 0 for each participant and counting participants with decrease in polyp burden at 12 months.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 15 | 19
Participants | 4 | 6
Statistical Analysis 1: Comparison: Arm I (Curcumin) vs Arm II (Placebo); Test type: Superiority; p = 0.85, Chi-squared

4. Secondary Outcome: Number of Participants With Grade >=2 Adverse Events
Description: Events were graded as follows:
  Grade 0= no adverse event or within normal limits; Grade 1= mild adverse event (causing no limitations of usual activity); Grade 2= moderate adverse event (causing some limitation of activity); Grade 3= severe adverse event (severe and undesirable; causing inability to carry out usual activities; Grade 4= life threatening or disabling adverse event; Grade 5= fatal adverse event.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 21 | 23
Participants | 6 | 2
Statistical Analysis 1: Comparison: Arm I (Curcumin) vs Arm II (Placebo); Test type: Superiority; p = 0.16, Chi-squared

5. Secondary Outcome: Medication Compliance
Description: Medication compliance of the participant= number of capsules taken divided by the number of capsules prescribed as determined by pill count and described as a percentage per participant. Then the compliance of each participant in the assigned group (curcumin or placebo) was averaged together to obtain the medication compliance rate of that group.
Time Frame: Up to 12 months
Measure: Median (Full Range); unit: percentage of total compliance
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 19 | 23
percentage of total compliance | 0.83 [0.70 to 0.94] | 0.91 [0.78 to 0.96]
Statistical Analysis 1: Comparison: Arm I (Curcumin) vs Arm II (Placebo); Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Ornithine Decarboxylase (ODC) Activity Levels
Description: Change in ODC mean activity levels (expressed as nmol of activity/mg of mucosal tissue/hr) at 8 months compared to baseline (time 0)
Time Frame: Baseline and 8 months
Measure: Mean (Standard Deviation); unit: nmol/mg/hr
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 21 | 23
nmol/mg/hr | 1.19 (0.71) | 0.88 (1.58)
Statistical Analysis 1: Comparison: Arm I (Curcumin) vs Arm II (Placebo); Test type: Superiority; p = 0.63, t-test, 2 sided

7. Secondary Outcome: Change in Total Polyamines Levels
Description: Polyamine mean level changes (expressed as pg/mg protein) at month 8-baseline
Time Frame: Baseline and 8 months
Measure: Mean (Standard Deviation); unit: pg/mg protein
Groups:
- Arm I (Curcumin): Patients receive curcumin PO BID for 12 months.
  Curcumin: Given PO
  Laboratory Biomarker Analysis: Correlative studies
- Arm II (Placebo): Patients receive placebo PO BID for 12 months.
  Laboratory Biomarker Analysis: Correlative studies
  Placebo: Given PO
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 21 | 23
pg/mg protein | 0.23 (3.41) | 1.66 (3.69)
Statistical Analysis 1: Comparison: Arm I (Curcumin) vs Arm II (Placebo); Test type: Superiority; p = 0.24, t-test, 2 sided

8. Secondary Outcome: Change in Micro RNA 124-U6 (miR124-U6)
Description: Change in MicroRNA mean activity level at 8 months compared to baseline (time 0)
Time Frame: Baseline and 8 months
Measure: Mean (Standard Deviation); unit: qRT-PCR relative to U6 snRNA
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 21 | 23
qRT-PCR relative to U6 snRNA | 1.44 (1.08) | 4.88 (11.55)
Statistical Analysis 1: Comparison: Arm I (Curcumin) vs Arm II (Placebo); Test type: Superiority; p = 0.63, t-test, 2 sided

9. Secondary Outcome: Change in Spermidine/Spermine N-1 Acetyl Transferase (SSAT)
Description: Change in SSAT mean activity level at 8 months compared to baseline (time 0)
Time Frame: Baseline and 8 months
Measure: Mean (Standard Deviation); unit: pmol/acetylspermidine/mg protein/min
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 21 | 23
pmol/acetylspermidine/mg protein/min | 0.97 (0.51) | 0.99 (0.56)
Statistical Analysis 1: Comparison: Arm I (Curcumin) vs Arm II (Placebo); Test type: Superiority; p = 0.93, t-test, 2 sided

10. Secondary Outcome: Change in Spermine Oxidase (SMOX)
Description: Change in SMOX mean activity level at 8 months compared to baseline (time 0)
Time Frame: Baseline and 8months
Measure: Mean (Standard Deviation); unit: pmol H2O2 per min per mg protein
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 21 | 23
pmol H2O2 per min per mg protein | 1.20 (0.57) | 1.56 (2.36)
Statistical Analysis 1: Comparison: Arm I (Curcumin) vs Arm II (Placebo); Test type: Superiority; p = 0.41, t-test, 2 sided

11. Secondary Outcome: Change in Ki-67 Anti-proliferative Cell Nuclear Antibody Index Levels
Description: Change in cellular proliferation rate was measured by assessment of Ki-67 anti-proliferative cell nuclear antibody index levels at 8 months
Time Frame: Baseline up to 8 months
Population: Specimens for analysis were only available on 7 curcumin and 10 placebo participants.
Measure: Mean (Standard Deviation); unit: labeled cells/crypt epithelial cells
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 7 | 10
labeled cells/crypt epithelial cells | 0.47 (0.21) | 0.41 (0.10)
Statistical Analysis 1: Comparison: Arm I (Curcumin) vs Arm II (Placebo); Test type: Superiority; p = 0.14, t-test, 2 sided

12. Secondary Outcome: Change in Apoptosis Index Levels
Description: Change in apoptosis index levels at 8 months by assessing cleaved Caspase-3 measurement
Time Frame: 8 months
Population: Specimens for analysis were only available on 7 curcumin and 10 placebo participants.
Measure: Mean (Standard Deviation); unit: apoptotic rate
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 7 | 10
apoptotic rate | 0.57 (0.98) | 2.44 (2.74)
Statistical Analysis 1: Comparison: Arm I (Curcumin) vs Arm II (Placebo); Test type: Superiority; p = 0.09, t-test, 2 sided

13. Other Pre Specified Outcome: Change in Mucosal DNA Methylation Levels.
Time Frame: Baseline to up to 12 months
Population: The outcome data were not collected and the outcome will never be analyzed.
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Change in Mucosal Leukotriene Levels.
Time Frame: Baseline to up to 12 months.
Population: The outcome data were not collected and the outcome will never be analyzed.
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

15. Other Pre Specified Outcome: Change in Mucosal Prostaglandin Levels.
Time Frame: Baseline to up to 12 months.
Population: The outcome data were not collected and the outcome will never be analyzed.
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

16. Other Pre Specified Outcome: Number of Patients Failing Study.
Description: Patients withdrawn from study due to increasing polyp burden and/or advancing histology.
Time Frame: Up to 16 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 21 | 23
Participants | 1 | 1
Statistical Analysis 1: Comparison: Arm I (Curcumin) vs Arm II (Placebo); Test type: Superiority; p = 0.95, Chi-squared

17. Other Pre Specified Outcome: Change in Vascular Density
Time Frame: Baseline up to 12 months
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

18. Other Pre Specified Outcome: Activation of NFKB (Nuclear Factor Kappa-light-chain-enhancer of Activated B Cells) Pathway
Time Frame: Baseline to 12 months
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

19. Other Pre Specified Outcome: Change in Akt Phosphorylation Levels
Time Frame: Baseline up to 12 months
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Reported adverse events (AE) included events starting on or after day 0 and on or before month 16.
Description: If a subject experienced more than 1 of a given AE the subject is counted only once for that AE. If a subject experienced more than 1 AE in a system organ class the subject is only counted once.
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/23
Serious Adverse Events (participants affected / at risk) | 3/21 | 1/23
Other Adverse Events (participants affected / at risk) | 8/21 | 13/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Curcumin) (N=21) | Arm II (Placebo) (N=23)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) — Subject developed appendicitis unrelated to study drug.
Facial abscess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Curcumin) (N=21) | Arm II (Placebo) (N=23)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Iron deficiency anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Herpes Zoster (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Headache migraine (Vascular disorders) | 0 (0) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Facial abscess (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Back strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar fascilitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Torn ligament (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less